CLINICAL TRIAL: NCT05123664
Title: A Prospective, Randomized, Placebo-controlled, Double-blind Study to Assess the Efficacy of Bacillus Coagulans Unique IS2 on Improving Bowel Movement Characteristics, Gastrointestinal-related Symptoms and Quality of Life in Healthy Adult Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2006
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Stool Frequency
Keywords: B. coagulans; probiotic; Bristol stool chart; GIQLI
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All capsules have the same appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacillus coagulans (Experimental): 2 billion CFU Bacillus coagulans Unique IS2 per capsule
  Interventions: Other: Capsule
- Placebo (Placebo Comparator): Appearance-matched capsule
  Interventions: Other: Capsule

INTERVENTIONS:
Other: Capsule — 1 cap daily at same time of the day with or without food for 4 weeks

SUMMARY:
This prospective, randomized, placebo-controlled, double-blind study will be conducted to assess the efficacy of 2 billion CFU/day of B. coagulans Unique IS2 on improving bowel movement characteristics, gastrointestinal-related symptoms and quality of life in healthy adult participants who are experiencing more than 3.0 but less than 6.0 complete spontaneous bowel movements (CSBM) per week on average.

Following a run-in period of 14 days to assess participants' baseline bowel habits, they are randomized to either B. coagulans or placebo for one month. The primary endpoint is change from baseline at 4 weeks in stool frequency in the test product group compared to the placebo group for average number of daily bowel movements over the week prior to the study visits. Secondary endpoints are stool frequency at weeks 1, 2, 3, stool quality measured by Bristol stool type scores, and gastrointestinal quality of life index (GIQLI) scores and subcategories (social, physical, emotional, symptoms).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adult participants who are 18 to 65 years of age (inclusive).
2. In good general health and good oral health (no active or uncontrolled diseases or conditions).
3. Have a body mass index (BMI) between 18.5 to 34.9 kg/m2 (inclusive).
4. Have normal (or acceptable to the investigator) vital signs (blood pressure and heart rate) at screening (Visit 1) and baseline (Visit 2) and normal (or acceptable to the investigator) physical exam findings (if applicable) at screening.
5. Individuals of childbearing potential must agree to practice a medically acceptable form of birth control for a defined timeframe prior to the start of run-in and throughout the study to avoid pregnancy, including:

   1. use for at least 3 months prior to run-in: hormonal contraceptives including oral contraceptives, hormone birth control patch (e.g., Ortho Evra), vaginal contraceptive ring (e.g., NuvaRing), injectable contraceptives (e.g., Depo-Provera, Lunelle), hormone implant (e.g., Norplant System), or intrauterine devices (e.g., Mirena); or
   2. use for at least 1 month prior to run-in: double-barrier method (e.g., condom with diaphragm or condom with cervical cap), non-hormonal intrauterine devices (i.e., copper), or complete abstinence from sexual intercourse that can result in pregnancy; or
   3. vasectomy of partner at least 6 months prior to run-in. Individuals with the potential to impregnate others must agree to avoid pregnancy by using the double-barrier method mentioned above or complete abstinence from sexual intercourse that can result in pregnancy.
6. Agree to refrain from treatments in the defined timeframes as outlined in Section 6.5.
7. Agree not to change current dietary habits (with the exception of avoiding pro- and prebiotic supplements), smoking and alcohol consumption habits, and activity/training levels starting from the beginning of the run-in period and for the duration of the study.
8. Agree to avoid anal penetration for 72 hours prior to fecal sample collection.
9. Agree to not receive a vaccine for COVID-19 throughout the duration of the study.
10. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.
11. At Visit 2/baseline, based on study diary data, an average of ≥3.0 and <7.0 weekly SBM (occurring without use of laxatives/suppositories/enema/manual maneuvers to defecate on the day of bowel movements or the day before) during the run-in period.
12. At Visit 2/baseline, achieve a study product compliance of 80-120% (inclusive) for the run-in period.

Exclusion criteria:

1. Participants who are lactating, pregnant or planning to become pregnant during the study.
2. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients, or not able to take any of the rescue medications.
3. Received a vaccine for COVID-19 in the last 2 weeks prior to screening, current COVID-19 infections, or COVID-19 long haulers (those who were first infected with COVID-19 ≥28 days prior to screening and continue to have symptoms).
4. Current diagnosis or history of irritable bowel syndrome (IBS), constipation (defined as an average of <3 defecations weekly for ≥3 months), inflammatory bowel disease (IBD, including ulcerative colitis and Crohn's disease), functional constipation or diarrhea (defined by the Rome IV diagnostic criteria), celiac disease, lactose intolerance and/or malabsorption, gastroparesis, gastroenteritis within the past 60 days, endometriosis, diverticulosis, gastric or duodenal ulcers, pancreatitis, or eating disorder; history of intestinal surgery (excluding appendectomy or herniorrhaphy), or history of bariatric surgery.
5. Constipation (defined as <3 defecations on average per week), and/or diarrhea (defined as ≥3 loose or liquid stools/day on any day) during run-in (based on daily diary at Visit 2/baseline).
6. Use of concomitant treatments within the defined timeframes as outlined in Section 6.5.
7. Change of dietary habits (e.g., starting a FODMAP diet, ketogenic diet or fiber supplement use, major increase or major decrease in consumption of high-fiber foods, etc.) within the 4 weeks prior to the beginning of the run-in period.
8. Having a history of heart disease, uncontrolled high blood pressure (≥140 systolic or ≥90 diastolic mmHg), renal or hepatic impairment/disease, uncontrolled diabetes (Type I or Type II), bipolar disorder, hepatic or renal dysfunction, unstable thyroid disease, immune disorders and/or immunocompromised (e.g. HIV/AIDS), a history of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit), or a history of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influence the results or the potential participant's ability to participate in the study.
9. Major surgery in 3 months prior to screening or planned major surgery during the course of the study.
10. History of alcohol or substance abuse, as deemed by the investigator, in the 12 months prior to screening.
11. Receipt or use of test product(s) in another research study within 30 days prior to run-in or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
12. Any other active or unstable medical conditions or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Stool frequency | Change from 7 day average prior to baseline versus 7 day average in fourth week. A significant increase is desirable.
  Number of daily bowel movements

SECONDARY OUTCOMES:
Stool frequency | Change from 7 day average prior to baseline to week 1, week 2 and week 3 averages. An increase from baseline stool frequency at Weeks 1, 2, or 3 in the B coagulans group, which is significantly better than the change in the placebo group, is desirable.
  Number of daily bowel movements
Stool quality | Change from 7 day average prior to baseline to week 1, 2, 3 and 4 average scores. An increase from baseline stool frequency in the B. coagulans group at weeks 1,2,3,4 which is significantly better than the change in the placebo group, is desirable.
  Bristol stool chart scale rated Type 1 (separate hard lumps) to Type 7 (watery, no solid pieces)
Gastrointestinal quality of life index | Change from baseline score to week 4 score. An improved score is desirable.
  Gastrointestinal quality of life index (GIQLI) total scores based on subcategory scores (social, physical, emotional, symptoms). 36 items are each rated from 0 (all the time) to 4 (never)

OTHER OUTCOMES:
Fecal microbiome composition | Shifts from baseline to Week 4. A better composition is desirable.
  Exploratory outcome: Microbial populations and their relative abundance assessed via 16S rRNA sequencing from fecal samples
Ratio of complete spontaneous bowel movements (SBMs) to total bowel movements | Changes from baseline to Week 4 in the test product group compared to the placebo group. More compete spontaneous bowel movements are better.
  The ratio of complete SBM to total bowel movements over one week will be multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.
Locations (1):
- Nutrasource Pharmaceutical and Nutraceutical Services, Inc.: Nutrasource Clinical Trial Site, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LeMoire A, Replogle R, Shinn L, Kamil A, Lin L, Kuttenkeuler AP, Baisley J, Wang J, Girard SA, Recker S, Bier A. Bacillus coagulans Unique IS2 improves stool characteristics in healthy adults with infrequent bowel movements: a randomized, double-blind, placebo-controlled trial. Benef Microbes. 2025 Jun 1;16(5):533-543. doi: 10.1163/18762891-bja00072. PMID 40456531